CLINICAL TRIAL: NCT02547662
Title: Phase 2 Trial of Pomalidomide, Ixazomib and Dexamethasone in Patients With Multiple Myeloma With Extramedullary Disease or Plasma Cell Leukemia
Brief Title: Pomalidomide, Ixazomib Citrate, and Dexamethasone in Treating Patients With Previously Treated Multiple Myeloma or Plasma Cell Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC1487; NCI-2015-01481 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2015-09-10; First posted 2015-09-11 (Estimated); Results first posted 2022-05-23 (Actual); Last update posted 2023-10-30 (Actual); Status verified 2023-10

CONDITIONS: Plasma Cell Leukemia; Plasma Cell Myeloma; Plasmacytoma
MeSH Terms: conditions — Leukemia, Plasma Cell; Multiple Myeloma; Plasmacytoma | interventions — Dexamethasone; Calcium Dobesilate; auricularum; dexamethasone acetate; dexamethasone 21-phosphate; ixazomib; pomalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (ixazomib citrate, pomalidomide, dexamethasone) (Experimental): Patients receive ixazomib citrate PO on days 1, 8, and 15, pomalidomide PO on days 1-21, and dexamethasone PO on days 1, 8, 15, and 22. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Dexamethasone; Drug: Ixazomib Citrate; Other: Laboratory Biomarker Analysis; Drug: Pomalidomide

INTERVENTIONS:
Drug: Dexamethasone — Given PO
  Other Names: Aacidexam; Adexone; Aknichthol Dexa; Alba-Dex; Alin; Alin Depot; Alin Oftalmico; Amplidermis; Anemul mono; Auricularum; Auxiloson; Baycuten; Baycuten N; Cortidexason; Cortisumman; Decacort; Decadrol; Decadron; Decalix; Decameth; Decasone R.p.; Dectancyl; Dekacort; Deltafluorene; Deronil; Desamethasone; Desameton; Dexa-Mamallet; Dexa-Rhinosan; Dexa-Scheroson; Dexa-sine; Dexacortal; Dexacortin; Dexafarma; Dexafluorene; Dexalocal; Dexamecortin; Dexameth; Dexamethasonum; Dexamonozon; Dexapos; Dexinoral; Dexone; Dinormon; Fluorodelta; Fortecortin; Gammacorten; Hexadecadrol; Hexadrol; Lokalison-F; Loverine; Methylfluorprednisolone; Millicorten; Mymethasone; Orgadrone; Spersadex; Visumetazone
Drug: Ixazomib Citrate — Given PO
  Other Names: MLN-9708; MLN9708; Ninlaro
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Pomalidomide — Given PO
  Other Names: 4-Aminothalidomide; Actimid; CC-4047; Imnovid; Pomalyst

SUMMARY:
This phase II trial studies how well pomalidomide, ixazomib citrate, and dexamethasone work in treating patients with previously treated multiple myeloma or plasma cell leukemia. Biological therapies, such as pomalidomide and dexamethasone, use substances made from living organisms that may stimulate or suppress the immune system in different ways and stop cancer cells from growing. Ixazomib citrate may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Giving pomalidomide, ixazomib citrate, and dexamethasone together may be more effective in treating multiple myeloma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the confirmed response rate (>= partial response [PR]) of ixazomib citrate (ixazomib), used in combination with pomalidomide and dexamethasone in patients with previously treated multiple myeloma (MM) with extramedullary disease.

SECONDARY OBJECTIVES:

I. To determine the toxicities associated with ixazomib in combination with pomalidomide and dexamethasone in patients with previously treated MM with extramedullary disease.

II. To determine the differential response rates (biochemical versus extramedullary disease) with ixazomib in combination with pomalidomide and dexamethasone in patients with previously treated MM with extramedullary disease.

III. To determine the progression free survival following treatment with ixazomib in combination with pomalidomide and dexamethasone in patients with previously treated MM with extramedullary disease.

TERTIARY OBJECTIVES:

I. To assess the proportion of patients achieving minimal residual disease (MRD) negative status.

OUTLINE:

Patients receive ixazomib citrate orally (PO) on days 1, 8, and 15, pomalidomide PO on days 1-21, and dexamethasone PO on days 1, 8, 15, and 22. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 or 6 months for up to 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Previously treated myeloma, currently with extramedullary disease (defined as plasmacytoma outside bone marrow that is not contiguous with a bone lesion) with at least one lesion that has a single diameter of >= 2 cm or plasma cell leukemia (defined as circulating plasma cells exceeding 5% of peripheral blood leukocytes or 0.5 X 10^9/L or 200 cells/150000 events by flow cytometry)
* Calculated creatinine clearance (using Cockcroft-Gault equation) >= 30 mL/min
* Absolute neutrophil count (ANC) >= 1000/mm^3
* Platelet count >= 50,000/mm^3
* Hemoglobin >= 8.0 g/dL
* Patients with measurable disease defined as at least one of the following:

  * For patients with extramedullary disease (EMD) measurable disease by computed tomography (CT) or magnetic resonance imaging (MRI) or the CT portion of the positron emission tomography (PET)/CT: must have at least one lesion that has a single diameter of >= 2 cm; skin lesions can be used if the area is >= 2 cm in at least one diameter and measured with a ruler
  * Plasma cell count >= 0.5 X 10^9/L or 5 percent of the peripheral blood white cells
  * Plasma cell count if determined by flow cytometry, >= 200/150,000 events
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0, 1 or 2
* Provide informed written consent
* Negative pregnancy test done =< 7 days prior to registration, for women of childbearing potential only
* All study participants must be registered into the mandatory pomalidomide (POMALYST) Risk Evaluation and Mitigation Strategy (REMS) program, and be willing and able to comply with the requirements of the POMALYST REMS program
* Willing to return to enrolling institution for follow-up (during the active monitoring phase of the study)
* Willing to provide bone marrow and blood samples for correlative research purposes

Exclusion Criteria:

* Other malignancy requiring active therapy

  * EXCEPTIONS: Non-melanoma skin cancer, ductal breast carcinoma in situ (DCIS) or carcinoma-in-situ of the cervix
  * NOTE: If there is a history or prior malignancy, they must not be receiving other specific treatment for their cancer
* Females of childbearing potential (FCBP)* must have a negative serum pregnancy test with a sensitivity of at least 50 mIU/mL within 10-14 days prior to and again within 24 hours prior to prescribing pomalidomide for cycle 1 (prescriptions must be filled within 7 days as required by RevAssist [lenalidomide REMS program]), and must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control, one highly effective method and one additional effective method; AT THE SAME TIME, at least 28 days before she starts taking pomalidomide FCBP must also agree to ongoing pregnancy testing; men must agree to use a latex condom during sexual contact with a FCBP even if they have had a successful vasectomy; patient must follow pregnancy testing requirements as outlined in the POMALYST REMS program

  * A female of childbearing potential is a sexually mature woman who: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months)
* Nursing women
* Men or women of childbearing potential who are unwilling to employ adequate contraception
* Other co-morbidity which would interfere with patient's ability to participate in trial, e.g. uncontrolled infection, uncompensated heart or lung disease
* Other concurrent chemotherapy, radiotherapy, or any ancillary therapy considered investigational

  * NOTE: Bisphosphonates are considered to be supportive care rather than therapy, and are thus allowed while on protocol treatment
* Patient has >= grade 3 peripheral neuropathy, or grade 2 with pain on clinical examination during the screening period
* Major surgery =< 14 days before study registration
* Systemic treatment with strong CYP3A4 inducers (e.g. rifampin, rifapentine, rifabutin, carbamazepine, phenytoin, phenobarbital, gingko biloba, St. John's wort) within 7 days before registration
* Evidence of current uncontrolled cardiovascular conditions, including cardiac arrhythmias, congestive heart failure, angina, or myocardial infarction within the past 6 months; Note: prior to study entry, any electrocardiogram (ECG) abnormality at screening must be documented by the investigator as not medically relevant
* Corrected QT Interval (QTc) > 470 milliseconds (msec) on a 12-lead ECG obtained during the screening period

  * Note: If a machine reading is above this value, the ECG should be reviewed by a qualified reader and confirmed on a subsequent ECG
* Known human immunodeficiency virus (HIV) positive
* Known hepatitis B surface antigen-positive status, or known or suspected active hepatitis C infection
* Any serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with the completion of treatment according to this protocol
* Known allergy to any of the study medications, their analogues or excipients in the various formulations
* Known gastrointestinal (GI) disease or GI procedure that could interfere with the oral absorption or tolerance of ixazomib including difficulty swallowing
* Diarrhea > grade 1, based on the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) grading, in the absence of antidiarrheals

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2015-12-24 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2020-10-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shaji Kumar, Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Mayo Clinic, Rochester, Minnesota
  - Sarah Cannon Cancer Center, Nashville, Tennessee

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study closed early due to recruitment concerns
Groups:
- Treatment (Ixazomib Citrate, Pomalidomide, Dexamethasone): Patients receive ixazomib citrate PO on days 1, 8, and 15, pomalidomide PO on days 1-21, and dexamethasone PO on days 1, 8, 15, and 22. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Dexamethasone: Given PO Ixazomib Citrate: Given PO Laboratory Biomarker Analysis: Correlative studies Pomalidomide: Given PO
Period: Overall Study
Arm/Group | Treatment (Ixazomib Citrate, Pomalidomide, Dexamethasone)
Started | 17
Completed | 17
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Ixazomib Citrate, Pomalidomide, Dexamethasone)
Number analyzed (Participants) | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.2 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 17
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 16
  More than one race | 0
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Confirmed Response Rate
Description: A confirmed response is defined as a patient who has achieved a stringent complete response (sCR), complete response (CR), very good partial response (PR), or PR on two consecutive evaluations. The proportion of successes will be estimated by the number of successes divided by the total number of evaluable patients. Ninety-five percent confidence intervals for the true success proportion will be calculated according to the approach of Duffy and Santner. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: 4 years
Measure: Number (95% Confidence Interval); unit: proportion of patients
Arm/Group | Treatment (Ixazomib Citrate, Pomalidomide, Dexamethasone)
Number analyzed (Participants) | 17
proportion of patients | 0.06 [0.0 to 0.29]

2. Secondary Outcome: Biochemical Response Rate
Description: The biochemical response rate will be estimated by the number of responders(patients that achieved partial or complete response) divided by the number of evaluable patients who have measurable disease by serum M-protein, urine M-protein, or serum FLC assay at baseline. Exact binomial confidence intervals will be calculated.
Time Frame: 4 years
Population: All patients evaluated for biochemical response
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Treatment (Ixazomib Citrate, Pomalidomide, Dexamethasone)
Number analyzed (Participants) | 12
proportion of participants | 0.25 [0.05 to 0.57]

3. Secondary Outcome: Extramedullary Response Rate
Description: Extramedullary response, defined as a response by extramedullary plasmacytoma or plasma cell count parameters. The extramedullary response rate will be estimated by the number of responders(patients that achieved a partial or complete response) divided by the number of evaluable patients. Exact binomial confidence intervals will be calculated.
Time Frame: 4 years
Population: All patients with extramedullary disease that were evaluated for response.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Treatment (Ixazomib Citrate, Pomalidomide, Dexamethasone)
Number analyzed (Participants) | 5
proportion of participants | 0.40 [0.05 to 0.85]

4. Secondary Outcome: Incidence of Adverse Events Graded According to the National Cancer Institute Common Terminology Criteria for Adverse Events Version 4.0
Description: Number of patients with adverse events is reported here, the full list of those adverse events and their frequency is reported in the adverse event section.
Time Frame: 4 years 1 month
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Ixazomib Citrate, Pomalidomide, Dexamethasone)
Number analyzed (Participants) | 17
Participants | 17

5. Secondary Outcome: Progression-free Survival
Description: The distribution of progression-free survival will be estimated using the method of Kaplan-Meier.
Time Frame: 4 years 8 months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment (Ixazomib Citrate, Pomalidomide, Dexamethasone)
Number analyzed (Participants) | 17
Months | 4.5 [2.0 to 11.8]

6. Other Pre Specified Outcome: Proportion of Patients Who Achieve Minimal Residual Disease (MRD) Negative Status
Description: The proportion of patients who achieve MRD negative status will be estimated by the number of patients who are MRD negative divided by the total number of evaluable patients who achieve a sCR or CR. Exact binomial 95% confidence intervals for the true MRD negative rate will be calculated.
Time Frame: Up to 5 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events were followed for 4 years and 1 month, mortality was followed for 4 years and 8 months.
Arm/Group | Treatment (Ixazomib Citrate, Pomalidomide, Dexamethasone)
All-Cause Mortality (participants affected / at risk) | 3/17
Serious Adverse Events (participants affected / at risk) | 5/17
Other Adverse Events (participants affected / at risk) | 17/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Ixazomib Citrate, Pomalidomide, Dexamethasone) (N=17)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Death NOS (General disorders) | 1 (1)
Infections and infestations - Oth spec (Infections and infestations) | 1 (1)
Lung infection (Infections and infestations) | 3 (4)
Upper respiratory infection (Infections and infestations) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Creatinine increased (Investigations) | 1 (1)
Lymphocyte count decreased (Investigations) | 1 (1)
Platelet count decreased (Investigations) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Neoplasms benign, mal, uncpec - Oth spec (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1)
Intracranial hemorrhage (Nervous system disorders) | 1 (1)
Confusion (Psychiatric disorders) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Ixazomib Citrate, Pomalidomide, Dexamethasone) (N=17)
Anemia (Blood and lymphatic system disorders) | 16 (47)
Eye disorders - Other, specify (Eye disorders) | 1 (6)
Constipation (Gastrointestinal disorders) | 10 (55)
Diarrhea (Gastrointestinal disorders) | 5 (6)
Nausea (Gastrointestinal disorders) | 9 (13)
Edema limbs (General disorders) | 2 (3)
Fatigue (General disorders) | 14 (102)
Pain (General disorders) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (4)
Creatinine increased (Investigations) | 7 (39)
Lymphocyte count decreased (Investigations) | 4 (7)
Neutrophil count decreased (Investigations) | 13 (40)
Platelet count decreased (Investigations) | 12 (41)
White blood cell decreased (Investigations) | 13 (30)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (4)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (2)
Peripheral motor neuropathy (Nervous system disorders) | 2 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 10 (79)
Tremor (Nervous system disorders) | 1 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2020-04-21): https://cdn.clinicaltrials.gov/large-docs/62/NCT02547662/Prot_SAP_ICF_000.pdf